CLINICAL TRIAL: NCT07287930
Title: The Safety and Efficacy of YTS109 Cell for Relapsed/Refractory Autoimmune Hemolytic Anemia Patients After Receiving Three or More Lines of Therapy.
Brief Title: A Study of YTS109 Cell in Subjects With Relapsed/Refractory Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS109-011
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: YTS109 cell (Experimental): Subjects will receive YTS109 cell, and dose escalation will commence at 1E6 cells/kg or the starting dose may be adjusted based on accumulated data.
  Interventions: Drug: YTS109 cell

INTERVENTIONS:
Drug: YTS109 cell — Subjects will receive YTS109 cell, and dose escalation will commence at 1E6 cells/kg or the starting dose may be adjusted based on accumulated data.

SUMMARY:
This is a Phase I, single-arm, open-label, dose-escalation and dose-expansion study. The primary objective is to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of YTS109 STAR-T cell therapy in patients with autoimmune hemolytic anemia who have failed ≥3 lines of therapy. The objective is to evaluate the safety, preliminary efficacy, pharmacokinetics/pharmacodynamics (PK/PD), and immune cell reconstitution characteristics of YTS109 cell therapy in Multi-rAIHA subjects who have failed third-line or higher-line treatments.

This study will also conduct an exploratory investigation into the impact of non-lymphodepleting conditioning prior to the infusion of STAR-T cells. For the non-lymphodepleting exploratory cell infusion, it can be administered as a single infusion or divided into 1 to 3 infusions (with the fractionated infusions to be completed within 7 days (and in any case no later than 15 days)). Dose escalation will commence at 1E6 cells/kg or the starting dose may be adjusted based on accumulated data.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, regardless of gender.
* A definitive diagnosis of Autoimmune Hemolytic Anemia (AIHA) or Evans Syndrome [including warm antibody-type, mixed warm-cold antibody-type, and cold antibody-type hemolytic anemia (cold agglutinin disease)] has been established, with diagnostic criteria referenced from the Chinese Clinical Practice Guidelines for the Diagnosis and Treatment of Autoimmune Hemolytic Anemia in Adults (2023 Edition).
* Patients who have undergone at least three failed treatment attempts, whose anemia symptoms (hemoglobin < 100 g/L) persist despite conventional therapy, and who remain unresponsive or experience recurrence after disease remission. Definition of Conventional Therapy: Treatment with glucocorticoids and/or rituximab, combined with any one or more of the following interventions: splenectomy, cyclosporine, cyclophosphamide, azathioprine, mycophenolate mofetil, bendamustine, fludarabine, bortezomib, or other pharmacological agents, as well as biologic agents including anti-CD38 monoclonal antibodies, BTK inhibitors, Syk inhibitors, complement inhibitors, etc.
* Adequate Organ Function:

  1. Liver Function:

     Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN); Total bilirubin ≤ 2.0 × ULN (excluding Gilbert syndrome, where total bilirubin ≤ 3.0 × ULN).
  2. Renal Function:

     Creatinine clearance (CrCl) ≥ 60 ml/minute (calculated using the Cockcroft-Gault formula).
  3. Oxygen Saturation (SpO₂): ≥ 92%.
  4. Bone Marrow Function Requirements:

     1. Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L;
     2. Platelet count ≥ 30 × 10⁹/L;
     3. International normalized ratio (INR) ≤ 1.5 × ULN;
     4. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
* ECOG performance status≤2.
* Subjects of childbearing potential will be required to follow contraception requirements from the time of enrollment until the end of the 12-month safety follow-up period.
* The subjects voluntarily participate in the study, sign the informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

* • Diagnosis of lymphoproliferative tumor

  * Other hereditary or acquired hemolytic diseases (Secondary AIHA caused by drugs or infection)
  * The platelet count in peripheral blood<30×10^9/L
  * Pregnant or breast-feeding subjects
  * Receive any of the following treatments within the specified time before cell infusion: a.anti-CD20 monoclonal antibodies <12 weeks, b.sutimlimab or other marketed biologics <5 half-lives,c.plasma exchange <4 weeks, d.post-splenectomy <12 weeks, e. BTK inhibitors, anti-CD38 monoclonal antibody, Syk inhibitors, BAFF inhibitors < 5 half-lives.
  * Previously received organ or stem cell transplantation
  * History of new thrombosis or organ infarction in the past 6 months
  * Diagnosis of the active stage of the connective tissue disease.
  * Have active infections, such as sepsis, bacteremia, fungemia, uncontrolled pulmonary infection and active tuberculosis, etc.
  * Positive hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg); positive hepatitis B e antibody (HBe-Ab) or hepatitis B core antibody (HBc-Ab), and the HBV-DNA copy number is above the lower limit of the measurable capacity; positive hepatitis C (HCV) antibody; positive human immunodeficiency virus (HIV) antibody; positive syphilis test.
  * Underwent major surgery within 4 weeks before screening, as determined by the investigator to be unsuitable for enrollment.
  * Have malignant tumors within 5 years before enrollment, except tumors with negligible risk of metastasis or death and curable tumors, such as adequately treated cervical carcinoma in situ, cutaneous basal cell carcinoma, etc.
  * Have any of the following cardiovascular diseases: a.Left ventricular ejection fraction (LVEF) ≤45%, b. presence of active heart disease or congestive heart failure (New York Heart Association [NYHA] Class III or IV)), c.severe arrhythmias requiring treatment, d.have myocardial infarction, bypass surgery, or stent placement within the 6 months before the study, e.other heart diseases judged by the researcher to be unsuitable for enrollment.
  * Have a history of live attenuated vaccines within 6 weeks before enrollment.
  * Have a history of epilepsy or other active central nervous system diseases.
  * Have an allergy to the ingredients of the medicine used in this study.
  * Previously received CAR-T cell therapy.
  * Patients considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
• Dose Limiting Toxicity [Time Frame: Within 28 days after infusion] | Within 28 days
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards.
• The incidence and frequency of treatment-emergent adverse events [Time Frame: Within 6 months after infusion] | Within 6 months
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards.

SECONDARY OUTCOMES:
• Best overall response rate (BOR) of each dose group [Time Frame: Within 12 weeks after infusion] | Within 12 weeks
  BOR is determined as the most favorable response observed after cell infusion, until either disease relapse or the completion of a specified observation
• Objective response rate (ORR) of each dose group [Time Frame: Within 4 weeks after infusion] | Within 4 weeks
• Time to response (TTR) [Time Frame: Within 6 months after infusion] | Within 6 months
  TTR is defined as the duration from cell infusion to the achievement of a hematological response
• Peak Plasma Concentration (Cmax) of YTS109 To evaluate the metabolic characteristics of YTS109 | Within 12 months after infusion
• Time to Peak (Tmax) of YTS109 To evaluate the metabolic characteristics of YTS109 | Within 12 months after infusion.
• Area under the plasma concentration versus time curve (AUC) of YTS109 To evaluate the metabolic characteristics of YTS109 | Within 12 months after infusion.
• The reconstitution of B cell in peripheral blood Changes in B cells quantification and phenotypic in peripheral blood | Within 12 months after infusion.

IPD SHARING:
Plan to Share IPD: No